CLINICAL TRIAL: NCT02951637
Title: Chemotherapy Plus Gefitinib Versus Gefitinib Alone as First-line Treatment for Patients With Advanced Lung Adenocarcinoma and Sensitive EGFR Mutations: a Randomized Controlled Trial
Brief Title: Chemotherapy Plus Gefitinib for Advanced Lung Adenocarcinoma and Sensitive EGFR Mutations: a Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Ruijin Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Aiqin Gu, Principal Investigator, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chest004
Record Dates: First submitted 2016-10-15; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Lung Adenocarcinoma
Keywords: Adenocarcinoma, EGFR, Gefitinib, Pemetrexed, Carboplatin
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma | interventions — Pemetrexed; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Patient will be administrated with Pemetrexed plus carboplatin combined with gefitinib
  Interventions: Drug: Pemetrexed plus carboplatin combined with gefitinib
- Group B (Experimental): Patient will be administrated with gefitinib
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Pemetrexed plus carboplatin combined with gefitinib — Pemetrexed (500mg/m(2) d1) plus carboplatin (AUC5 d1) combined with gefitinib (250mg d4-28) and repeat every four weeks for up to six cycles and then continue to receive pemetrexed combined with gefitinib every four weeks.
  Other Names: Combination of chemotherapy and EGFR TKI
  Arms: Group A
Drug: Gefitinib — Gefitinib (250mg daily)
  Other Names: EGFR TKI
  Arms: Group B

SUMMARY:
The purpose of this study is to compare chemotherapy and gefitinib in combination with gefitinib alone as first-line therapy for adenocarcinoma, in terms of efficacy and safety.

DETAILED DESCRIPTION:
The primary endpoints is to compare the progression-free survival (PFS) of pemetrexed plus carboplatin combined with gefitinib to gefitinib alone as first-line therapy for lung adenocarcinoma.

In addition, the overall survival and safety index will be collected for analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had to voluntarily join the study and give written informed consent for the study;
2. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC);
3. A cytologic diagnosis is acceptable (FNA or pleural fluid cytology)
4. Sensitive EGFR mutations (19del, 21L858R);
5. At least 1 unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST) criteria;
6. Patients did not receive systemic anti-cancer therapy previously;
7. Able to comply with study and follow-up procedures;
8. Age >= 18 years, ECOG PS: 0-1, estimated survival duration more than 3 months;

Exclusion Criteria:

1. Small cell lung cancer (including patients with mixed small cell lung cancer and non-small cell lung cancer);
2. Evidence of small cell, carcinoid, or mixed small cell/non-small cell histology;
3. EGFR wild-type patients, or patients with rare EGFR mutations or complex EGFR mutations;
4. Previously (within 5 years) or presently suffering from other malignancies, except for cured cervical carcinoma in situ, non-melanoma skin cancers and superficial bladder cancer [Ta (noninvasive carcinoma), Tis (carcinoma in situ) and T1 (invasion into lamina propria)];
5. Symptomatic or untreated brain metastases;
6. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or serious cardiac arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible);
7. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications;
8. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption;
9. Pregnancy or lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 16 months

SECONDARY OUTCOMES:
overall survival (OS) | 32 months
Objective response rate (ORR) | 6 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aiqin Gu, MD, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: Undecided